CLINICAL TRIAL: NCT03710356
Title: Essai Bayésien de Phase I/II évaluant l'efficacité et la tolérance du Danazol Chez Les Patients Ayant Une Atteinte hématologique ou Pulmonaire sévère liée à Une téloméropathie - ANDROTELO
Brief Title: Evaluating Efficacy and Safety of Danazol in Severe Hematologic or Pulmonary Disease Related to Telomeropathy
Acronym: ANDROTELO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170925J; 2018-001686-17 (EudraCT Number)
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Telomere Shortening; Telomere Length, Mean Leukocyte
MeSH Terms: interventions — Danazol

STUDY DESIGN:
Intervention Model Description: phase ½ therapeutic trial stratified on disease (Severe Hematologic or Pulmonary Disease)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Danazol (Experimental): Danazol
  Interventions: Drug: Danazol 200 MG

INTERVENTIONS:
Drug: Danazol 200 MG — DANAZOL 200 mg as capsules 800 mg/d orally, in 2 doses Duration of treatment: 12 months

SUMMARY:
Constitutional mutations of genes involved in telomere repair and maintenance are responsible for "telomeropathy" (" Congenital Dyskeratosis "). Attrition of telomeres promotes cell senescence and genetic instability. The penetrance and severity of organ damage (pulmonary, hematological, liver, and neurological) is variable, depending on the gene involved, the generation concerned (anticipation phenomenon) and also environmental factors.

In cases of bone marrow failure, the only curative treatment is hematopoietic stem cell transplant, often limited by pulmonary and / or hepatic involvement or the absence of a suitable HLA match donor. The pulmonary phenotype is most often that of idiopathic pulmonary fibrosis. In severe forms, a lung transplant is proposed in the absence of contraindications. Anti-fibrotic treatments are not very effective or not evaluated. The observed decrease in the vital capacity of these patients is 300 ml / year, abnormally high compared to idiopathic forms. Evolution without transplant is in both situations rapidly unfavorable; the prognosis after lung or marrow transplant is also worse than that of similar transplants without telomeres disease.

Danazol has been used for over 4 decades in acquired and constitutional bone marrow failure in the absence of a therapeutic alternative. In telomeropathy, retrospective data on small cohorts indicate a haematological response rate of 60-70%. A prospective study in the United States recently showed a haematological response at 1 year in 78% of cases (10 of 12 evaluable patients) with stabilization of vital capacity. Retrospective data (unpublished) on patients treated in France have shown more side effects and more frequent treatment interruptions and eventually weaker haematological response rate. This study aim to evaluate the benefit of danazol at 12 months on the clinical response.

ELIGIBILITY:
Inclusion Criteria:

* with telomeropathy defined by the existence of a deleterious constitutional mutation of a gene involved in telomere maintenance (TERT, TERC, DKC1, TINF2, RTEL1, PARN, ACD, NHP2, NOP10, NAF1, WRAP53, CTC1, ERCC6L2, USB1, POT1, DNAJC21 or a newly identified gene responsible for telomeropathy ),
* 15 years or older,
* with severe haematological involvement (platelets < 20 G/L or ANC < 0.5 G/L and/or hemoglobin < 8 g/dL and/or transfusion needs) and/or pulmonary fibrosis with parenchymal involvement greater than 10% on the CT scan.
* being able to give informed consent for patients 18 years and older,
* being able to give consent and have the consent of the holder (s) of parental authority for children over 15 years,
* being a beneficiary of social security scheme.

Exclusion Criteria:

* with HIV infection or active hepatitis B or C infection,
* with severe hepatic disease: ASAT and/or ALAT > 5N, or direct bilirubinemia > 30 μmol/L, TP <50% (except vitamin K deficiency),
* having an active or treated tumor pathology for less than 5 years with the exception of a basocellular carcinoma or a in situ carcinoma of the cervix,
* with a history of organ or hematopoietic stem cell transplantation or with an indication of hematopoietic stem cell or organ transplantation within 6 months of inclusion,
* with an absolute contraindication to treatment with danazol: active thrombosis or history of thromboembolic disease, porphyria, severe renal or cardiac insufficiency (NYHA stage III or IV), androgen-dependent tumor, uncharacterized mammary nodules, pathological genital hemorrhage of undetermined etiology,
* who have already received danazol for the treatment of telomeropathy,
* having received another androgen within a period of less than 6 months,
* receiving another experimental treatment,
* receiving another hormonal therapy,
* receiving simvastatin,
* having a pregnancy plan and not committing to effective contraception while taking the treatment,
* breastfeeding,
* under guardianship or curators.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2021-10-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Hematological response or Pulmonary response at M12 | 12 months
  Response at 12 months is defined according to the initial pathology. Responses is defined as a composite outcome. At least one of the following item should be validated to observe response.
  * For patients with bone marrow failure, the hematological response at 12 months depending on initial cytopenia(s) is defined by
  * 1.5 g/dL increase in hemoglobin without transfusion for 2 months
  * And/or increase of 20.10^9/L in platelet count without transfusion for 2 months
  * And/or increase of 0.5.10^9/L in neutrophils count.
  * For patients with pulmonary fibrosis, a decrease of less than 5% in forced vital capacity at 12 months

SECONDARY OUTCOMES:
Hepatic tolerance M1 | 1 month
  aspartate aminotransferase blood level
Hepatic tolerance M2 | 2 months
  aspartate aminotransferase blood level
Hepatic tolerance M3 | 3 months
  aspartate aminotransferase blood level
Hepatic tolerance M6 | 6 months
  aspartate aminotransferase blood level
Hepatic tolerance M9 | 9 months
  aspartate aminotransferase blood level
Hepatic tolerance M12 | 12 months
  aspartate aminotransferase blood level
LDL cholesterol M3 | 3 months
  Low-density lipoprotein (LDL) cholesterol blood level in mmol/l
LDL cholesterol M6 | 6 months
  Low-density lipoprotein (LDL) cholesterol blood level in mmol/l
LDL cholesterol M9 | 9 months
  Low-density lipoprotein (LDL) cholesterol blood level in mmol/l
LDL cholesterol M12 | 12 months
  Low-density lipoprotein (LDL) cholesterol blood level in mmol/l
HDL cholesterol M3 | 3 months
  High-density lipoprotein (LDL) cholesterol blood level in mmol/l
HDL cholesterol M6 | 6 months
  High-density lipoprotein (LDL) cholesterol blood level in mmol/l
HDL cholesterol M9 | 9 months
  High-density lipoprotein (LDL) cholesterol blood level in mmol/l
HDL cholesterol M12 | 12 months
  High-density lipoprotein (LDL) cholesterol blood level in mmol/l
TG M3 | 3 months
  triglycerides blood level in mmol/l
TG M6 | 6 months
  triglycerides blood level in mmol/l
TG M9 | 9 months
  triglycerides blood level in mmol/l
TG M12 | 12 months
  triglycerides blood level in mmol/l
PSA M3 | 3 months
  Prostate-specific antigen (PSA) blood level for men
PSA M6 | 6 months
  Prostate-specific antigen (PSA) blood level for men
PSA M12 | 12 months
  Prostate-specific antigen (PSA) blood level for men
Pulmonary parenchymal abnormalities M6 | 6 months
  Evolution of pulmonary parenchymal abnormalities at CT scan
Pulmonary parenchymal abnormalities M12 | 12 months
  Evolution of pulmonary parenchymal abnormalities at CT scan
Telomere length | 12 months
  Evolution of the telomere length by Flow Fish
cytological and cytogenetic abnormalities | 12 months
  Appearance of cytological and cytogenetic abnormalities (bone marrow aspiration with cytogenetic)
Quality of life evaluation M3 | 3 months
  European Organisation for Research and Treatment of Cancer Quality of Life of Cancer Patients questionnaire (EORTC QLQ-C30, v3.0). The scale range from to 30 to 126 (30 represents the worse quality of life and 126 the best quality of life).
  http://www.eortc.be/qol/files/C30/QLQ-C30%20English.pdf
Quality of life evaluation M6 | 6 months
  European Organisation for Research and Treatment of Cancer Quality of Life of Cancer Patients questionnaire (EORTC QLQ-C30, v3.0). The scale range from to 30 to 126 (30 represents the worse quality of life and 126 the best quality of life).
  http://www.eortc.be/qol/files/C30/QLQ-C30%20English.pdf
Quality of life evaluation M12 | 12 months
  European Organisation for Research and Treatment of Cancer Quality of Life of Cancer Patients questionnaire (EORTC QLQ-C30, v3.0). The scale range from to 30 to 126 (30 represents the worse quality of life and 126 the best quality of life).
  http://www.eortc.be/qol/files/C30/QLQ-C30%20English.pdf
Overall survival | 12 months
DLCO M3 | 3 months
  Diffusing capacity of the lung for carbon monoxide (DLCO)
DLCO M6 | 6 months
  Diffusing capacity of the lung for carbon monoxide (DLCO)
DLCO M9 | 9 months
  Diffusing capacity of the lung for carbon monoxide (DLCO)
DLCO M12 | 12 months
  Diffusing capacity of the lung for carbon monoxide (DLCO)

IPD SHARING:
Plan to Share IPD: No